CLINICAL TRIAL: NCT02510027
Title: Molecular Triage in Cervical Cancer Prevention: The Tlaxcala Study
Brief Title: Triage Strategies in Cervical Cancer Prevention
Acronym: FRIDA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Secretaria de Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Eduardo Cesar Lazcano Ponce, Eduardo Lazcano-Ponce, MD, DSc, Instituto Nacional de Salud Publica, Mexico
Other Study IDs: 1094
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Cervical Cancer; Intraepithelial Neoplasia
Keywords: HPV testing; Triage; Mexico; Cervical cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Carcinoma in Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two cervical samples will be collected using a Cervex-Brush® (Rovers®). The first collected sample will be placed in a vial containing BD CytoRich™ preservative (BD Diagnostics, Burlington, NC), and the second sample will be placed in a ThinPrep® vial (Hologic, Inc., Bedford, MA). Both samples will be temporarily stored at room temperature at the health center until they are delivered to the lab facilities. Women who refuse a pelvic examination will be offered the option to self-collect a vaginal sample at the health facility or at their home that can be used for hrHPV testing. Only HR-HPV positive participants will move onto the cytology/molecular triage testing phase. After triage procedures, all remaining samples collected in either of the vials from HR-HPV positive women will be stored independently for additional analysis as required by the study procedures.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women aged 30-64 years old: Women aged 30 to 64 years who attend the Cervical Cancer Screening Program in 100 health centers in the state of Tlaxcala, Mexico
  Interventions: Other: HPV screening and triage tests

INTERVENTIONS:
Other: HPV screening and triage tests — All cervical and/or vaginal specimens are tested for hrHPV using the Cobas® 4800 HPV test. Triage testing will be performed on all participants with a positive HR-HPV test declared consent at recruitment visit: HPV16/18 genotyping, Cobas® 4800 HPV test, HPV16/18/45 genotyping, BD OnclarityTM HPV Assay, OncoE6 Cervical Test, Liquid based cytology with Papanicolaou stain and p16INK4a/ Ki-67 immunostain.

SUMMARY:
While there is broad consensus that HR-HPV detection is the best available primary screening test, there is no agreement about the most efficient and reliable triage procedure for HR-HPV positive women. Transient HR-HPV infections are very common, and the vast majority of these infections spontaneously regress after a year or two. Only a small fraction of cases will lead to persistent infection responsible for cervical neoplasia. The FRIDA Study is a large, population-based study that was designed to evaluate the performance and cost-effectiveness of different triage strategies for hrHPV-positive women in Mexico.

DETAILED DESCRIPTION:
The target population is over <100,000 women aged 30 to 64 years who attend the Cervical Cancer Screening Program in 100 health centers in the state of Tlaxcala, Mexico. All women will be evaluated to determine hrHPV infection using the Cobas® 4800 HPV test. Triage strategies will be performed as reflex tests in all hrHPV-positive participants: HPV-16/18/45 genotyping, detection of the E6 oncoprotein of HPV-16/18, cytology, and immunocytochemistry using p16INK4a/Ki67. Women with at least one positive triage test will be referred for colposcopy evaluation, where a minimum of four biopsies and an endocervical sample are systematically collected. Histological confirmation will be performed by a standardized panel of pathologists.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30 to 64
* Residents of the municipalities included in Sanitary Jurisdiction No. 1 of Tlaxcala.

Exclusion Criteria:

* Pregnant or hysterectomized women
* Legally disabled women unable to give verbal informed consent required by the study protocol
* Women who do not wish to participate in the present study

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a population-based study that includes all women aged 30 to 64 years living in the 32 municipalities in Tlaxcala covered by Sanitary Jurisdiction No. 1 of Tlaxcala Health Services
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Histologically confirmed cervical intraepithelial neoplasia grade 2 or worse (CIN2+) | 36 months
  All women will be colposcopically evaluated in order to rule out any clinically evident invasive cancer. In cases of invasive cancer, patients will be referred to onco-gynecology services immediately. Before biopsy collection, endocervical sampling is performed using an Endocervex Brush®. A minimum of four biopsies are collected, at least one per quadrant, from the more suspicious area on cervical transformation zone. Histological evaluation of all samples (biopsies and/or endocervical curettage samples) will be evaluated for final diagnosis and confirmation of CIN2+ cases by two pathologists according to Mexico's Cervical Cancer Screening Programme's guidelines. An external expert-pathologist, will resolve discrepancies and render a final decision.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo C Lazcano-Ponce, MD DSc, Principal Investigator — Instituto Nacional de Salud Publica, Mexico
Locations (1):
- Primary health care centers from Sanitary Jurisdiction No. 1 of Tlaxcala Health Services, Tlaxcala City, Tlaxcala, Mexico

REFERENCES:
- [Derived] Torres-Ibarra L, Lorincz AT, Wheeler CM, Cuzick J, Hernandez-Lopez R, Spiegelman D, Leon-Maldonado L, Rivera-Paredez B, Mendez-Hernandez P, Lazcano-Ponce E, Salmeron J. Adjunctive testing by cytology, p16/Ki-67 dual-stained cytology or HPV16/18 E6 oncoprotein for the management of HPV16/18 screen-positive women. Int J Cancer. 2021 May 1;148(9):2264-2273. doi: 10.1002/ijc.33414. Epub 2020 Dec 22. PMID 33252834
- [Derived] Hernandez-Lopez R, Lorincz AT, Torres-Ibarra L, Reuter C, Scibior-Bentkowska D, Warman R, Nedjai B, Mendiola-Pastrana I, Leon-Maldonado L, Rivera-Paredez B, Ramirez-Palacios P, Lazcano-Ponce E, Cuzick J, Salmeron J; FRIDA Study Group. Methylation estimates the risk of precancer in HPV-infected women with discrepant results between cytology and HPV16/18 genotyping. Clin Epigenetics. 2019 Oct 12;11(1):140. doi: 10.1186/s13148-019-0743-9. PMID 31606044
- [Derived] Rudolph SE, Lorincz A, Wheeler CM, Gravitt P, Lazcano-Ponce E, Torres-Ibarra L, Leon-Maldonado L, Ramirez P, Rivera B, Hernandez R, Franco EL, Cuzick J, Mendez-Hernandez P, Salmeron J; FRIDA Study Group. Population-based prevalence of cervical infection with human papillomavirus genotypes 16 and 18 and other high risk types in Tlaxcala, Mexico. BMC Infect Dis. 2016 Sep 1;16(1):461. doi: 10.1186/s12879-016-1782-x. PMID 27585544